CLINICAL TRIAL: NCT02198937
Title: Investigation on the Effect of Smoking on the Expression of Pro- and Anti-thrombotic, Anti-oxidative, and Inflammatory Markers in Humans
Status: Terminated | Type: Observational
Why Stopped: Funding unclear
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Simon Staempfli, MD, University of Zurich
Other Study IDs: KEK-ZH-NR. 2014-0078
Record Dates: First submitted 2014-07-21; First posted 2014-07-24 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Inflammation; Thrombosis; Smoking
Keywords: smokers; non-smokers
MeSH Terms: conditions — Inflammation; Thrombosis; Smoking | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Blood sample

GROUPS / COHORTS (2):
- Smokers: Healthy smokers
  Interventions: Other: Blood sample
- Non-Smokers: Healthy non-smokers
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample

SUMMARY:
Investigation on the effect of smoking on thrombus formation in humans. The expression of pro- and anti-thrombotic, anti-oxidative, and inflammatory markers will be assessed in 25-50 year old healthy smokers and non-smokers. The investigators are interested in possible differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Smoker
* Non-smokers

Exclusion Criteria:

* Disease
* Pregnancy

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Smokers and non-smokers
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Expression of pro- and anti-thrombotic, anti-oxidative, and inflammatory markers in blood | Single time point, no follow-up (cross sectional)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Zurich, Switzerland